CLINICAL TRIAL: NCT06724926
Title: A Phase IB Study to Assess Safety of Concurrent Azeliragon With Craniospinal Irradiation in Patients With Leptomeningeal Metastasis From Solid Tumor Malignancies or High-Grade Gliomas
Brief Title: Concurrent Azeliragon With Craniospinal Irradiation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-00982
Record Dates: First submitted 2024-12-06; First posted 2024-12-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; High-grade Glioma; Leptomeningeal Metastasis
MeSH Terms: conditions — Glioma; Meningeal Carcinomatosis | interventions — azeliragon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Determination followed by Dose Expansion (Experimental): Patients with leptomeningeal metastasis from a solid tumor or primary CNS high-grade glioma will be enrolled and start Azeliragon 7 days prior to CSI, during CSI, and for 7 days days after completion of CSI (Dose Determination). Patients will be monitored for dose limiting toxicities during protocol therapy.
  Once the recommended dose is identified, additional patients will be treated with Azeliragon at recommended dose in combination with craniospinal irradiation (Dose Expansion).
  Interventions: Drug: Azeliragon; Procedure: CSI

INTERVENTIONS:
Drug: Azeliragon — Azeliragon is orally administered. Patients start Azeliragon 7 days before CSI and take their last dose 7 days post-CSI.
  The first 6 patients will start at Dose Level 1 [DL1] (Loading dose for 7 days: 30 mg twice daily; Concurrent/adjuvant dose: 20 mg once daily).
  If 1 or fewer of 6 patients develop dose-limiting toxicity (DLT) then the recommended dose will be DL1. If at least 2 of 6 develops a DLT, then an additional 6 patients will be enrolled at Dose Level -1 [DL-1] (Loading dose for 7 days: 15mg twice daily; Concurrent/adjuvant dose: 10mg once daily).
  If 1 or fewer out of 6 patients at DL-1 develop DLT, then the recommended dose will be DL-1. If at least 2 of 6 at DL-1 develops a DLT, then an additional 6 patients will be enrolled at Dose Level -2 [DL-2] (Loading dose for 7 days: 15mg twice daily; Concurrent/adjuvant dose: 5mg once daily).
  At the recommended dose, an additional 14 patients will be enrolled for the Dose Expansion portion.
Procedure: CSI — Patients will receive CSI.

SUMMARY:
Single institution study to assess the safety of concurrent Azeliragon with craniospinal irradiation (CSI) in patients with leptomeningeal metastasis from solid tumor malignancies and high-grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Patient with solid tumor malignancy or high grade glioma with leptomeningeal metastasis established radiographically and/or through cerebrospinal fluid (CSF) cytology
* Patients who are candidates for radiation therapy for the treatment of leptomeningeal metastasis
* Patients with Karnofsky Performance Status of 60 or greater.
* Male or non-pregnant and non-lactating female and ≥ 18 years of age.
* Patients with absolute neutrophil count (ANC) ≥ 1.0 × 109/L, platelet count ≥ 75,000/mm3 (75 × 109/L), and hemoglobin (Hgb) ≥ 8 g/dL. Transfusion or growth factor support is allowed.
* Patients with aspartate aminotransferase (AST) [serum glutamic-oxaloacetic transaminase(SGOT)], alanine aminotransferase (ALT) [serum glutamic-pyruvic transaminase (SGPT)] ≤ 2.5 × upper limit of normal range (ULN), unless liver metastases are present, then ≤ 5 x ULN is acceptable, total bilirubin ≤ 1.5 × ULN, and estimated creatinine clearance of > 30 mL/min (per Cockroft-Gault formula).
* Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria:

* Patient has a life expectancy, per investigator assessment, of less than 2 months.
* Patients unable to complete the English quality of life questionnaires
* Patient with extensive systemic disease and who declined standard systemic treatment options
* Patient who is unable to undergo magnetic resonance imaging (MRI) brain and spine with gadolinium contrast
* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerance
* Active, uncontrolled bacterial, or fungal infection(s) requiring systemic therapy.
* Patient has a concomitant serious medical or psychiatric illness that, in the opinion of the investigator, could compromise the patient's safety or the study data integrity.
* Patient is unwilling or unable to comply with study procedures, including, but not limited to self-administration of oral medication.
* Patients with a gastrointestinal condition that could interfere with swallowing or absorption.
* Females of childbearing potential who are sexually active or males with female partners of childbearing potential, where either the female or the male is unwilling to use a highly effective method of contraception during the trial and for 6 months after the last administration of study drug.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose-Limiting Toxicities (DLTs) at Dose Level 1 | Up to Week 4
  DLTs assess using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.
Number of Patients with DLTs at Dose Level -1 | Up to Week 4
  DLTs assess using CTCAE v 5.0.
Number of Patients with DLTs at Dose Level -2 | Up to Week 4
  DLTs assess using CTCAE v 5.0.

SECONDARY OUTCOMES:
Central nervous system (CNS) progression-free survival (PFS) | Up to Month 13 (12 Months Post-Protocol Therapy)
  CNS PFS is defined as time from randomization until CNS progression or death, whichever occurs first.
Overall Survival (OS) | Up to Month 13 (12 Months Post-Protocol Therapy)
  OS is defined as time from randomization until death.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Yang, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Jonathan.Yang@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Jonathan.Yang@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.